CLINICAL TRIAL: NCT02919995
Title: A Phase IIa, Randomised, Double Blind, Placebo Controlled, Three Way Crossover Study to Assess the Pharmacokinetics of RPL554 Administered to Adult Patients With Cystic Fibrosis.
Brief Title: A Study of RPL554 in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Collaborators: Cystic Fibrosis Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RPL554-010-2015; 2015-004263-36 (EudraCT Number)
Record Dates: First submitted 2016-09-21; First posted 2016-09-30 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2019-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ensifentrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Higher Dose RPL554 (Experimental): Single dose of inhaled 6 mg RPL554
  Interventions: Drug: RPL554
- Lower dose RPL554 (Experimental): Single dose of inhaled 1.5 mg RPL554
  Interventions: Drug: RPL554
- Placebo (Placebo Comparator): Inhaled placebo dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPL554 — RPL554 suspension administered using a nebuliser
  Arms: Higher Dose RPL554; Lower dose RPL554
Drug: Placebo — Placebo solution administered using a nebuliser
  Arms: Placebo

SUMMARY:
This study evaluates two doses of RPL554 and placebo in adult patients with cystic fibrosis. All patients receive all three treatments in a randomised sequence.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.

  2. Male or female aged ≥18 years at the time of informed consent. Females of childbearing potential must have been using a consistent and reliable form of contraception (see Appendix 1) from the last menses before the first study treatment administration, and must commit to continue to do so during the study and for 3 months after the last dose of study treatment.

  3. Have a 12-lead ECG recording at screening (Visit 1) and Visit 2 pre-dose showing the following:
  * Heart rate between 45 and 90 beats per minute
  * QT interval corrected for heart rate using Fridericia's formula (QTcF) interval ≤450 msec
  * QRS interval ≤120 msec
  * PR interval ≤220 msec
  * No clinically significant abnormality including morphology (e.g. left bundle branch block, atrioventricular nodal dysfunction, ST segment abnormalities) 4. Capable of complying with all study restrictions and procedures including ability to use the study nebuliser correctly.

    5. Body mass index (BMI) between 18 and 30 kg/m2 (inclusive) with a minimum weight of 40 kg.

    6. Patients with a genetic diagnosis of CF. 7. Spirometry at screening demonstrating an FEV1 ≥40% and ≤80% of predicted normal.

    8. Capable of withdrawing from long acting bronchodilators1 until the end of the treatment period, and short acting bronchodilators for 8 hours prior to administration of study treatment.

    9. Clinically stable CF in the 2 weeks prior to randomisation (Visit 2).

Exclusion Criteria:

1. History of cirrhotic liver disease or portal hypertension.
2. CF exacerbation requiring hospitalisation in the month prior to screening (Visit 1) or prior to randomisation (Visit 2).
3. Use of oral or intravenous antibiotics (in additional to usual maintenance therapy) in the 2 weeks prior to screening (Visit 1) or randomisation (Visit 2).
4. Other non-CF related respiratory disorders: Patients with a current diagnosis of active tuberculosis, lung cancer, sarcoidosis, sleep apnoea, known alpha-1 antitrypsin deficiency or other active pulmonary diseases.
5. Previous lung resection or lung transplant.
6. History of, or reason to believe a patient has, drug or alcohol abuse within the past 3 years.
7. Received an experimental drug within 3 months or five half-lives, whichever is longer.
8. Patients with a history of chronic uncontrolled disease including, but not limited to, cardiovascular (including arrhythmias), endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, haematological, urological, immunological or ophthalmic diseases that the Investigator believes are clinically significant.
9. Documented cardiovascular disease: angina, recent or suspected myocardial infarction, congestive heart failure, a history of unstable, or uncontrolled hypertension, or has been diagnosed with hypertension in last 3 months.
10. Has had major surgery, (requiring general anaesthesia) in the 6 weeks prior to screening (Visit 1) or will not have fully recovered from surgery, or planned surgery through the end of the study.
11. Infection with nontuberculous mycobacteria, methicillin-resistant Staphylococcus aureus (MRSA), or Burkholderia species.
12. Use of immune-suppression; long term use of prednisolone ≥10 mg/day.
13. History of malignancy of any organ system within 5 years with the exception of localised skin cancers (basal or squamous cell).
14. Clinically significant abnormal values for safety laboratory tests (haematology, biochemistry or urinalysis) at screening (Visit 1), as determined by the Investigator.
15. A disclosed history or one known to the Investigator, of significant non-compliance in previous investigational studies or with prescribed medications.
16. Requires oxygen therapy, even on an occasional basis.
17. Pregnancy or lactation (female subjects only).
18. Any other reason that the Investigator considers makes the patient unsuitable to participate. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Floto, Principal Investigator — Cambridge Centre for Medical Research, Papworth Hospital
Locations (1):
- Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 patients were screened; six patients failed screening. Patients had to discontinue long acting bronchodilators on the day prior to screening and short acting bronchodilators for 8 hours before all spirometry assessments
Groups:
- Higher Dose RPL554/Lower Dose RPL554/Placebo: Single dose of inhaled 6 mg RPL554 in Period 1, Single inhaled dose of 1.5 mg RPL554 in Period 2, placebo in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Lower Dose RPL554/Placebo/Higher Dose RPL554: Single dose of inhaled 1.5 mg RPL554 in Period 1, single inhaled dose of placebo in Period 2, single inhaled dose of 6 mg RPL554 in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Higher Dose RPL554/Plaebo/Lower Dose RPL554: Single inhaled dose of 6 mg RPL554 in Period 1, single inhaled dose of placebo in Period 2, single inhaled dose of 1.5 mg RPL554 in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Lower Dose RPL554/Higher Dose RPL554/Placebo: Single inhaled dose of 1.5 mg RPL554 in Period 1, single inhaled dose of 6 mg RPL554 in Period 2, single inhaled dose of placebo in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Placebo/Higher Dose RPL554/Lower Dose RPL554: Single inhaled dose of placebo in Period 1, single inhaled dose of 6 mg RPL554 in Period 2, single inhaled dose of 1.5 mg RPL554 in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Placebo/Lower Dose RPL554/Higher Dose RPL554: Single inhaled dose of placebo in Period 1, single inhaled dose of 1.5 mg RPL554 in Period 2, single inhaled dose of 6 mg RPL554 in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
Period: Overall Study
Arm/Group | Higher Dose RPL554/Lower Dose RPL554/Placebo | Lower Dose RPL554/Placebo/Higher Dose RPL554 | Higher Dose RPL554/Plaebo/Lower Dose RPL554 | Lower Dose RPL554/Higher Dose RPL554/Placebo | Placebo/Higher Dose RPL554/Lower Dose RPL554 | Placebo/Lower Dose RPL554/Higher Dose RPL554
Started | 1 | 2 | 2 | 2 | 1 | 2
Completed | 1 | 2 | 2 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Higher Dose RPL554/Lower Dose RPL554/Placebo: Single dose of inhaled 6 mg RPL554 in Period 1, single dose of inhaled 1.5 mg RPL554 in Period 2, single inhaled dose of placebo in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Lower Dose RPL554/Placebo/Higher Dose RPL554: Single dose of inhaled 1.5 mg RPL554 in Period 1, single dose of inhaled placebo RPL554 in Period 2, single dose of 6 mg RPL554 in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Higher Dose RPL554/Placebo/Lower Dose RPL554: Single dose of inhaled 6 mg RPL554 in Period 1, single dose of inhaled placebo in Period 2, single dose of inhaled 1.5 mg RPL554 in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Lower Dose RPL554/Higher Dose RPL554/Placebo: Single dose of inhaled 1.5 mg RPL554 in Period 1, single dose of inhaled 6 mg RPL554 in Period 2, single inhaled dose of placebo in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Placebo/Higher Dose RPL554/Lower Dose RPL554: Single dose of inhaled placebo in Period 1, single dose of inhaled 6 mg RPL554 in Period 2, single dose of inhaled 1.5 mg RPL554 in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Placebo/Lower Dose RPL554/Higher Dose RPL554: Single dose of inhaled placebo in Period 1, single dose of inhaled 1.5 mg RPL554 in Period 2, single dose of inhaled 6 mg RPL554 in Period 3
  RPL554: RPL554 suspension administered using a nebuliser Placebo: Placebo solution administered using a nebuliser
- Total: Total of all reporting groups
Arm/Group | Higher Dose RPL554/Lower Dose RPL554/Placebo | Lower Dose RPL554/Placebo/Higher Dose RPL554 | Higher Dose RPL554/Placebo/Lower Dose RPL554 | Lower Dose RPL554/Higher Dose RPL554/Placebo | Placebo/Higher Dose RPL554/Lower Dose RPL554 | Placebo/Lower Dose RPL554/Higher Dose RPL554 | Total
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 1 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 2 | 1 | 2 | 10
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 1 | 0 | 1 | 4
  Male | 1 | 2 | 0 | 1 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 2 | 2 | 1 | 2 | 10
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC by Dose
Description: Area under the curve (AUC)
Time Frame: Pre dose, 15 and 30 minutes and 1, 2, 4, 6, 8 and 24 hours post dose after each treatment
Population: All randomised patients with blood sampling performed after at least one dose of RPL554 and with data sufficient to calculate pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Higher Dose RPL554 | Lower Dose RPL554
Number analyzed (Participants) | 9 | 9
pg*h/mL | 7699 (2965.7) | 2342 (1029.9)

2. Primary Outcome: Maximum Plasma Concentration After Each Dose
Description: Maximum plasma concentration (Cmax) after a single dose of RPL554
Time Frame: Pre dose, 15 and 30 minutes and 1, 2, 4, 6, 8 and 24 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Higher Dose RPL554 | Lower Dose RPL554
Number analyzed (Participants) | 9 | 9
pg/mL | 828.3 (256.1) | 270.1 (91.9)

3. Primary Outcome: Time to Maximum Plasma Concentration After Each Dose
Description: Time to maximum concentration (Tmax) after a single dose of RPL554
Time Frame: Pre dose, 15 and 30 minutes and 1, 2, 4, 6, 8 and 24 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Higher Dose RPL554 | Lower Dose RPL554
Number analyzed (Participants) | 9 | 9
hours | 1.53 (0.66) | 1.33 (0.62)

4. Primary Outcome: Half Life for Each Dose
Description: Half life (t1/2) of RPL554
Time Frame: Pre dose, 15 and 30 minutes and 1, 2, 4, 6, 8 and 24 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Higher Dose RPL554 | Lower Dose RPL554
Number analyzed (Participants) | 9 | 9
Hours | 10.14 (3.1) | 7.52 (3.3)

5. Secondary Outcome: Peak FEV1 for Each Treatment
Description: Maximum Forced expired volume in one second (FEV1) measured using spirometry
Time Frame: Pre dose and 15 and 30 minutes and 1, 2 and 4 hours post dose after treatment
Population: All randomized patients with sufficient data collected after intake of study treatment to compute the pharmacodynamic parameters on at least two study visits.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Higher Dose RPL554 | Lower Dose RPL554 | Placebo
Number analyzed (Participants) | 9 | 10 | 10
Liters | 2.384 (0.73) | 2.247 (0.72) | 2.256 (0.71)
Statistical Analysis 1: Comparison: Lower Dose RPL554 vs Placebo; Test type: Other; p = 0.0196, ANCOVA; Contrast ratio = 1.038, 95% CI 2-sided [1.007 to 1.07]
Statistical Analysis 2: Comparison: Higher Dose RPL554 vs Placebo; Test type: Other; p = 0.0802, ANCOVA; Contrast ratio = 1.024, 95% CI 2-sided [0.997 to 1.052]
Statistical Analysis 3: Comparison: Higher Dose RPL554 vs Lower Dose RPL554; Test type: Other; p = 0.3487, ANCOVA; Contrast ratio = 0.986, 95% CI 2-sided [0.957 to 1.017]

6. Secondary Outcome: AUC FEV1(0-4h)
Description: Area under the curve for FEV1 over 4 hours measured using spirometry
Time Frame: Pre dose and 15 and 30 minutes and 1, 2 and 4 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Higher Dose RPL554 | Lower Dose RPL554 | Placebo
Number analyzed (Participants) | 9 | 10 | 10
Liters | 2.313 (0.73) | 2.194 (0.72) | 2.133 (0.73)
Statistical Analysis 1: Comparison: Lower Dose RPL554 vs Placebo; Test type: Other; p = 0.0043, ANCOVA; Contrast ratio = 1.072, 95% CI 2-sided [1.026 to 1.12]
Statistical Analysis 2: Comparison: Higher Dose RPL554 vs Placebo; Test type: Other; p = 0.0109, ANCOVA; Contrast ratio = 1.055, 95% CI 2-sided [1.014 to 1.096]
Statistical Analysis 3: Comparison: Higher Dose RPL554 vs Lower Dose RPL554; Test type: Other; p = 0.4306, ANCOVA; Contrast ratio = 0.984, 95% CI 2-sided [0.942 to 1.027]

7. Secondary Outcome: AUC FEV1(0-6h)
Description: Area under the curve FEV1 over 6 hours measured using spirometry
Time Frame: Pre dose and 15 and 30 minutes and 1, 2, 4 and 6 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Higher Dose RPL554 | Lower Dose RPL554 | Placebo
Number analyzed (Participants) | 9 | 10 | 10
Liters | 2.304 (0.74) | 2.188 (0.73) | 2.133 (0.73)
Statistical Analysis 1: Comparison: Lower Dose RPL554 vs Placebo; Test type: Other; p = 0.0064, ANCOVA; Contrast ratio = 1.065, 95% CI 2-sided [1.021 to 1.11]
Statistical Analysis 2: Comparison: Higher Dose RPL554 vs Placebo; Test type: Other; p = 0.0149, ANCOVA; Contrast ratio = 1.049, 95% CI 2-sided [1.011 to 1.089]
Statistical Analysis 3: Comparison: Higher Dose RPL554 vs Lower Dose RPL554; Test type: Other; p = 0.466, ANCOVA; Contrast ratio = 0.945, 95% CI 2-sided [0.945 to 1.027]

8. Secondary Outcome: AUC FEV1(0-8h)
Description: Area under the curve for FEV1 over 8 hours measured using spirometry
Time Frame: pre dose and 15 and 30 minutes and 1, 2, 4, 6 and 8 hours post dose
Population: All randomised patients with sufficient data collected after intake of study treatment to compute the pharmacodynamic parameters on at least two study visits.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Higher Dose RPL554 | Lower Dose RPL554 | Placebo
Number analyzed (Participants) | 9 | 10 | 10
Liters | 2.287 (0.75) | 2.185 (0.74) | 2.130 (0.74)
Statistical Analysis 1: Comparison: Lower Dose RPL554 vs Placebo; Test type: Other; p = 0.0093, ANCOVA; Contrast ratio = 1.061, 95% CI 2-sided [1.017 to 1.107]
Statistical Analysis 2: Comparison: Higher Dose RPL554 vs Placebo; Test type: Other; p = 0.0333, ANCOVA; Contrast ratio = 1.042, 95% CI 2-sided [1.004 to 1.082]
Statistical Analysis 3: Comparison: Higher Dose RPL554 vs Lower Dose RPL554; Test type: Other; p = 0.3693, ANCOVA; Contrast ratio = 0.982, 95% CI 2-sided [0.941 to 1.024]

9. Secondary Outcome: FVC
Description: Forced vital capacity (FVC) measured using spirometry
Time Frame: Over 24 hours after treatment
Reporting Status: Not Posted

10. Secondary Outcome: Breath Samples
Description: Exhaled breath pH
Time Frame: 8 and 24 hours after treatment
Reporting Status: Not Posted

11. Secondary Outcome: Laboratory Safety Tests 1
Description: Biochemistry panel parameters
Time Frame: Screening and end of study
Reporting Status: Not Posted

12. Secondary Outcome: Laboratory Safety Tests 2
Description: Haematology panel parameters
Time Frame: Screening and end of study
Reporting Status: Not Posted

13. Secondary Outcome: Laboratory Safety Tests 3
Description: Urinalysis measured by urine dipstick
Time Frame: Screening and end of study
Reporting Status: Not Posted

14. Secondary Outcome: Vital Signs 1
Description: Pulse rate after 5 minutes supine
Time Frame: Over 8 hours after treatment
Reporting Status: Not Posted

15. Secondary Outcome: Vital Signs 2
Description: Blood pressure after 5 minutes supine
Time Frame: Over 8 hours after treatment
Reporting Status: Not Posted

16. Secondary Outcome: ECG 1
Description: Heart rate
Time Frame: Over 8 hours after treatment
Reporting Status: Not Posted

17. Secondary Outcome: ECG 2
Description: QT interval
Time Frame: Over 8 hours after treatment
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Sputum Rheology
Description: Rheological analysis for interleukin 8, tumour necrosis factor alpha and myeloperoxidase
Time Frame: 8 and 12 hours after treatment
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Sputum Measurements
Description: Levels of inflammatory mediators
Time Frame: 8 and 12 hours after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From informed consent through study completion, up to 52 days
Arm/Group | Higher Dose RPL554 | Lower Dose RPL554 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/9 | 6/10 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher Dose RPL554 (N=9) | Lower Dose RPL554 (N=10) | Placebo (N=10)
exacerbation of cystic fibrosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher Dose RPL554 (N=9) | Lower Dose RPL554 (N=10) | Placebo (N=10)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of cystic fibrosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall not be permitted to present at symposia, national or regional professional meetings, nor publish in journals, theses or dissertations, or otherwise of their own choosing, methods and results of the Clinical Trial without the prior written approval of the Sponsor. Any such approved presentation or publication shall acknowledge the Sponsor as the sponsor of the Clinical Trial and owner of the results of the Clinical Trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT02919995/Prot_002.pdf
  • Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT02919995/SAP_000.pdf